CLINICAL TRIAL: NCT05842967
Title: A PHASE 3 PROTOCOL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS (RSV) PREFUSION F SUBUNIT VACCINE IN ADULTS AT HIGH RISK OF SEVERE RSV DISEASE
Brief Title: A Study to Assess the Safety, Tolerability, and Immunogenicity of RSVpreF in Adults at High Risk of Severe RSV Disease
Acronym: MONET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C3671023; NCT05842967 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: RESPIRATORY SYNCYTIAL VIRUS (RSV)
Keywords: RESPIRATORY SYNCYTIAL VIRUS (RSV); ADULTS AT HIGH RISK; IMMUNOCOMPROMISED ADULTS

STUDY DESIGN:
Intervention Model Description: Substudy A: Phase 3, multicenter, randomized, double-blinded, placebo-controlled study that will assess the safety, tolerability, and immunogenicity of Pfizer's RSVpreF in adults 18 to <60 years of age considered to be at high risk of RSV disease due to certain chronic medical conditions. Approximately 675 participants ≥18 to <60 years of age considered at high risk of RSV disease due to certain chronic medical conditions, excluding immunocompromising conditions, will be randomized to receive a single 120-µg dose of RSVpreF or placebo in a 2:1 ratio.
  Substudy B: Phase 3, single-arm, open-label, multicenter study that will assess the safety, tolerability, and immunogenicity of Pfizer's RSVpreF in immunocompromised adults. Approximately 200 immunocompromised adults ≥18 years of age will receive 2 120-µg doses of RSVpreF with an interval of 1 month. Approximately 100 participants will be ≥60 years of age and approximately 100 participants will be ≥18 to 60 years of age.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Substudy A is double blind therefore all parties (participant, site staff and sponsor) will be blinded to study intervention.
  Substudy B is open-label therefore no blinding requirements are in place since all participants will receive RSVpreF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Substudy A - RSVpreF (Experimental): Participants will receive a single 120-µg dose of RSVpreF at Visit 1
  Interventions: Biological: RSVpreF
- Substudy A - Placebo (Placebo Comparator): Participants will receive placebo at Visit 1
  Interventions: Other: Placebo
- Substudy B - RSVpreF (Experimental): Participants will receive 120-µg doses of RSVpreF at Visit 1 and Visit 2 (open label, single arm only)
  Interventions: Biological: RSVpreF

INTERVENTIONS:
Biological: RSVpreF — 120-µg
  Arms: Substudy A - RSVpreF; Substudy B - RSVpreF
Other: Placebo — Placebo
  Arms: Substudy A - Placebo

SUMMARY:
The purpose of this study is to learn about the safety and immunogenicity of a study vaccine (called RSVpreF) in several adult groups. Respiratory Syncytial Virus (RSV) is a common type of virus (germ) that can cause severe illness, where medical help is needed. RSV can lead to airway diseases in all ages. Vaccines help your body make antibodies which help fight against diseases. This is called an immune response. This study will measure how much antibody participants make after receiving RSVpreF (immunogenicity).

The study consists of 2 groups (Substudy A and Substudy B).

Substudy A is seeking approximately 675 participants who are:

* Between 18 and 60 years of age.
* Considered having a high likelihood of severe RSV disease due to certain long-term medical conditions. Such medical conditions do not include immunocompromising conditions.

Participants will need to come to the study clinic at least 2 times. At the first clinic visit, participants will receive 1 shot of RSVpreF or placebo in the arm by chance. A placebo looks like the study vaccine but contains no active ingredients. At each clinic visit, a blood sample will be taken. A third (final) visit can be either completed in clinic or via telephone contact. This study is about 6 months long for each participant.

Substudy B is seeking approximately 200 participants who are:

* At least 18 years of age. About half of the participants will be at least 60 years of age.
* Considered having a weakened immune system (immunocompromised). Participants will need to come to the study clinic at least 3 times. All participants will receive a shot of RSVpreF at the first study clinic visit. The second study clinic visit will be 1 month later. All participants will receive a second shot of the study vaccine at this second study clinic visit. Blood samples will be taken at the 3 study clinic visits. A fourth (final) visit can be either completed in clinic or via telephone contact. This study is about 7 months long for each participant.

DETAILED DESCRIPTION:
This is a Phase 3 protocol that will assess the safety, tolerability, and immunogenicity of Pfizer's RSVpreF in adults at high risk of severe RSV disease. Each substudy design is detailed separately, and these substudies may be conducted in parallel, as required by the clinical plan, within the framework of this protocol.

Substudy A Design:

This is a Phase 3, multicenter, randomized, double-blinded, placebo-controlled study that will assess the safety, tolerability, and immunogenicity of Pfizer's RSVpreF in adults 18 to <60 years of age considered to be at high risk of RSV disease due to certain chronic medical conditions.

Approximately 675 participants ≥18 to <60 years of age considered at high risk of RSV disease due to certain chronic medical conditions, excluding immunocompromising conditions, will be randomized to receive a single 120-µg dose of RSVpreF or placebo in a 2:1 ratio. Enrollment will be monitored to help ensure distribution of vaccination across the age range. The duration of study participation for each participant will be 6 months, with 3 scheduled visits.

All participants will have blood drawn at baseline prior to vaccination and at 1 month after vaccination to assess immunogenicity. Immunogenicity elicited at 1 month after vaccination with RSVpreF in Substudy A will be bridged to the immunogenicity of participants 60 years of age and older in the C3671013 study, in which RSVpreF efficacy was demonstrated.

Local reaction and systemic event data will be collected in an e-diary for 7 days after study vaccination (Days 1 through 7, where Day 1 is the day of vaccination). Reported Grade 3 reactogenicity will be assessed by the study site to determine if an unscheduled visit is required.

For all participants, AEs will be collected from informed consent through 1 month following study intervention administration, and AESIs, NDCMCs and SAEs will be collected from informed consent throughout study participation. In addition, AEs occurring up to 48 hours after blood draws that are related to study procedures will be collected.

Substudy B Design:

This is a Phase 3, single-arm, open-label, multicenter study that will assess the safety, tolerability, and immunogenicity of Pfizer's RSVpreF in immunocompromised adults.

Substudy B included approximately 200 immunocompromised adults ≥18 years of age, that will receive 2 120-µg doses of RSVpreF with an interval of 1 month. Approximately 100 participants will be ≥60 years of age and approximately 100 participants will be ≥18 to 60 years of age. Enrollment will be monitored to help ensure distribution of vaccination across the age ranges and underlying immunocompromising conditions. The duration of study participation for each participant will be 7 months, with 4 scheduled visits. All participants will have blood drawn at baseline prior to vaccination and at 1 month after (each) vaccination to assess immunogenicity.

Local reaction and systemic event data will be collected in an e-diary for 7 days after study vaccination (Days 1 through 7, where Day 1 is the day of vaccination). Reported Grade 3 reactogenicity will be assessed by the study site to determine if an unscheduled visit is required.

For all participants, AEs will be collected from informed consent through 1 month following the last study intervention administration, and AESIs, NDCMCs and SAEs will be collected from informed consent throughout study participation. In addition, AEs occurring up to 48 hours after blood draws that are related to study procedures will be collected.

ELIGIBILITY:
Substudy A Inclusion Criteria:

1. Capable of giving signed informed consent as described per protocol.
2. Participants ≥18 to <60 years of age at study enrollment.
3. Life expectancy ≥12 months (365 days) in the opinion of the investigator at enrollment.
4. Participants who are willing and able to comply with all scheduled visits, vaccination plan, lifestyle considerations, and other study procedures.
5. Participants who are considered at high risk of RSV disease by virtue of the following:

   * Adults with chronic pulmonary (including asthma), cardiovascular (excluding isolated hypertension), renal, hepatic, neurologic, hematologic, or metabolic disorders (including diabetes mellitus).

Chronic medical conditions for this substudy are defined as:

- Duration greater than 6 months.

* Stable disease not requiring a significant change in therapy in the previous 6 weeks or hospitalization for worsening disease within 12 weeks before receipt of study intervention.
* Requires regular medical follow-up or ongoing medication or hospitalization in the previous year.

  • Additional groups at high risk include:
* Residents of nursing homes and other long-term care facilities.

Substudy A Exclusion Criteria:

1. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
2. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s) or any related vaccine.
3. Participants who do not have adequate deltoid muscle mass to allow intramuscular vaccination, in the opinion of the investigator.
4. Serious chronic disorder, including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
5. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Note: Specific criteria for participants with known stable infection with HIV can be found in protocol.
7. Individuals who receive chronic systemic treatment with immunosuppressive therapy, including cytotoxic agents, immunosuppressive monoclonal antibodies, systemic corticosteroids*, eg, for cancer or an autoimmune disease, or radiotherapy, from 60 days before study intervention administration or planned receipt throughout the study.

   *Applies to systemic corticosteroids administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent (eg, for cancer or an autoimmune disease). Systemic corticosteroids administered at a dose of <20 mg/day of prednisone or equivalent are permitted. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin, eyes, or ears) corticosteroids are permitted.
8. Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration or planned receipt of these medications prior to the final blood draw.

   Note: Monoclonal antibodies with targeted mechanisms of action used in the management of chronic illnesses (eg, migraine headaches, osteoporosis) are permitted, provided they do not meet exclusion criterion 7.
9. Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.
10. Participation in other studies involving an investigational product within 28 days prior to consent and/or through and including the 6-month follow-up visit.
11. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Substudy B Inclusion Criteria

1. Capable of giving signed informed consent as described per protocol.
2. Participants ≥18 years of age at study enrollment.
3. Life expectancy ≥12 months (365 days) in the opinion of the investigator at enrollment.
4. Participants who are willing and able to comply with all scheduled visits, vaccination plan, lifestyle considerations, and other study procedures.
5. Participants who are immunocompromised by virtue of the following:

   •Having known advanced NSCLC with at least 1 of the following:
   * Has received initial or maintenance chemotherapy at least 2 weeks (14 days) before enrollment (or is treatment-naïve), and is not expected to receive chemotherapy within at least 2 weeks (14 days) after dose administration of initial vaccination or second vaccination; and/or
   * Is receiving checkpoint inhibitor treatment (PD-1/PD-L1 inhibitor, CTLA-4 inhibitor) and has undergone at least 1 treatment cycle prior to enrollment; or
   * Is receiving targeted drug therapy (EGFR, ALK, ROS1, BRAF, RET, MET, NTRK inhibitors) and has undergone at least 1 treatment cycle prior to enrollment.

   OR - Is currently undergoing maintenance hemodialysis treatment secondary to end-stage renal disease . OR - Is on active immunomodulator therapy (eg, TNFα inhibitor, tofacitinib, or MTX) for an autoimmune inflammatory disorder (eg, inflammatory arthritis, such as rheumatoid arthritis, psoriatic arthritis, and juvenile idiopathic arthritis, or inflammatory bowel disease, such as ulcerative colitis or Crohn's disease) at a stable*dose.

   *Stable dose is defined as receiving the same dose for at least 3 months (84 days) with no changes in the 28 days prior to enrollment. See protocol for details on stable dose for MTX.

   OR - Is receiving an SOT (kidney, liver, lung, or heart) at least 3 months (84 days) prior to enrollment (Visit 201) and with no acute rejection episodes within 2 months (60 days) prior to enrollment (Visit 201).

   Substudy B Exclusion Criteria:

1.Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.

2.History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s) or any related vaccine.

3.Participants with a history of transplant rejection, or PTLD, or participants who have had treatment for these conditions within 3 months (84 days) prior to study enrollment.

4.Participants who do not have adequate deltoid muscle mass to allow intramuscular vaccination, in the opinion of the investigator.

5.Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Note: Specific criteria for participants with known stable infection with HIV can be found in protocol.

6.Receipt of investigational or approved monoclonal antibodies against RSV within 6 months before study intervention administration.

7.Receipt of blood/plasma products or immunoglobulin (IVIG, SCIG) within 60 days before study intervention administration or planned receipt of these medications prior to the final blood draw.

Note: Please see the inclusion criteria in the protocol regarding criteria for targeted immunoglobulin therapies for underlying medical conditions.

Note: Monoclonal antibodies with targeted mechanisms of action used in the management of chronic illnesses (eg, migraine headaches, osteoporosis) are permitted.

8.Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.

9.Participation in other studies involving an investigational product within 28 days prior to consent and/or through and including the 6-month follow-up visit.

10.Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (36):
  - North Alabama Research Center, Athens, Alabama
  - Central Research Associates, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Hope Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Hope Research Institute, Tempe, Arizona
  - Orange County Research Center, Lake Forest, California
  - Kaiser Permanente, Los Angeles, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - GW Vaccine Research Unit, Washington D.C., District of Columbia
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Clinical Neuroscience Solutions - Orlando - South Delaney Avenue, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Institute of Human Virology (IHV), Baltimore, Maryland
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinical Applications LLC dba QPS-MO (Patient Screening Only), Springfield, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Wilmington, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Orion Clinical Research, Austin, Texas
  - AIM Trials, LLC, Plano, Texas
  - Epic Medical Research, Red Oak, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Almeida NC, Parameswaran L, DeHaan EN, Wyper H, Rahman F, Jiang Q, Li W, Patton M, Lino MM, Majid-Mahomed Z, Malkin E, Davis M, Towner WJ, Saharia K, Ilangovan K, Kalinina E, Cooper D, Swanson KA, Anderson AS, Gurtman A, Munjal I. Immunogenicity and Safety of the Bivalent Respiratory Syncytial Virus Prefusion F Subunit Vaccine in Immunocompromised or Renally Impaired Adults. Vaccines (Basel). 2025 Mar 19;13(3):328. doi: 10.3390/vaccines13030328. PMID 40266222
- [Derived] Davis M, Towner W, DeHaan E, Jiang Q, Li W, Rahman F, Patton M, Wyper H, Lino MM, Sarwar UN, Majid-Mahomed Z, Mehta S, Howitt W, Cannon K, Kalinina E, Cooper D, Swanson KA, Anderson AS, Gurtman A, Munjal I; MONeT Study Team. Bivalent RSVpreF Vaccine in Adults 18 to <60 Years Old With High-Risk Conditions. Clin Infect Dis. 2025 Apr 30;80(4):911-920. doi: 10.1093/cid/ciae550. PMID 39523547
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Substudy A (SSA) and substudy B (SSB) are reported differently. SSA was randomized; SSB was open-label single-arm. Enrollment number 885 derived from participants with IP assigned in SSA (681 randomized) and SSB (204). Since no randomization in SSB (single arm), tables of SSB present 217 participants as starting substudy (signed informed consent), out of which 203 vaccinated. In SSA: 678 vaccinated.
Pre-assignment Details: For immunogenicity analysis for SSA, as planned, data of participants >=60 years vaccinated with RSVpreF in C3671013 [NCT05035212] study is used for comparison. These participants were not enrolled in the present study C3671023 [NCT05842967], only the relevant historical data was used for comparison as per the objectives.
Groups:
- SSA: RSVpreF: Participants aged >=18 to <60 years received respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF) 120 microgram (mcg) intramuscularly on Day 1 of SSA.
- SSA: Placebo: Participants aged >=18 to <60 years received placebo (lyophile matched to RSVpreF) intramuscularly on Day 1 of SSA.
- SSB: RSVpreF, >= 18 to < 60 Years: Participants aged >=18 to <60 years received RSVpreF 120 mcg intramuscularly first dose on Day 1 of SSB (Vaccination 1) and second dose on 1-month post-vaccination 1 (Vaccination 2).
- SSB: RSVpreF, >= 60 Years: Participants aged >=60 years received RSVpreF 120 mcg intramuscularly first dose on Day 1 of SSB (Vaccination 1) and second dose on 1-month post-vaccination 1 (Vaccination 2).
Period: Period 1: SSA
Arm/Group | SSA: RSVpreF | SSA: Placebo | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Started | 454 | 227 | 0 | 0
Vaccinated | 453 | 225 | 0 | 0
Completed | 432 | 218 | 0 | 0
Not Completed | 22 | 9 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 4 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Not completed — Randomized but not vaccinated | 1 | 2 | 0 | 0
Period: Period 2: SSB
Arm/Group | SSA: RSVpreF | SSA: Placebo | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Started | 0 | 0 | 101 | 116
Vaccinated | 0 | 0 | 96 | 107
Completed | 0 | 0 | 89 | 103
Not Completed | 0 | 0 | 12 | 13
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Enrolled but not vaccinated | 0 | 0 | 5 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received the study intervention.
Groups:
- SSA: RSVpreF: Participants aged >=18 to <60 years received RSVpreF 120 mcg intramuscularly on Day 1 of SSA.
- Total: Total of all reporting groups
Arm/Group | SSA: RSVpreF | SSA: Placebo | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years | Total
Number analyzed (Participants) | 453 | 225 | 96 | 107 | 881
Age, Customized [Count of Participants; unit: Participants]
  18 to <60 years | 453 | 225 | 96 | 0 | 774
  >=60 years | 0 | 0 | 0 | 107 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260 | 152 | 56 | 53 | 521
  Male | 193 | 73 | 40 | 54 | 360
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 102 | 48 | 8 | 3 | 161
  Not Hispanic or Latino | 348 | 175 | 88 | 101 | 712
  Unknown or Not Reported | 3 | 2 | 0 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 3 | 5
  Asian | 24 | 9 | 6 | 2 | 41
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 0 | 4
  Black or African American | 106 | 57 | 25 | 15 | 203
  White | 312 | 152 | 63 | 87 | 614
  More than one race | 3 | 1 | 0 | 0 | 4
  Unknown or Not Reported | 5 | 5 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: SSA: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: Local reactions included pain at injection site, redness and swelling, recorded by participants in an electronic diary (e-diary). Pain at injection site was graded as mild: did not interfere with activity; moderate: interfered with activity and severe: prevented daily activity. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild: >2.5 cm to 5.0 cm; moderate: >5.0 cm to 10.0 cm; severe: >10 cm.
Time Frame: Within 7 Days after Vaccination (Vaccination on Day 1)
Population: E-diary safety population included all participants who received the study intervention with at least 1 day of e-diary data transmitted.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | SSA: RSVpreF | SSA: Placebo
Number analyzed (Participants) | 451 | 225
Percentage of Participants
  Pain at injection site: Mild | 29.7 [25.5 to 34.2] | 10.2 [6.6 to 14.9]
  Pain at injection site: Moderate | 5.5 [3.6 to 8.1] | 0.4 [0.0 to 2.5]
  Pain at injection site: Severe | 0 [0.0 to 0.8] | 0 [0.0 to 1.6]
  Redness: Mild | 3.8 [2.2 to 6.0] | 0 [0.0 to 1.6]
  Redness: Moderate | 2.2 [1.1 to 4.0] | 0.4 [0.0 to 2.5]
  Redness: Severe | 0 [0.0 to 0.8] | 0 [0.0 to 1.6]
  Swelling: Mild | 4.0 [2.4 to 6.2] | 0.4 [0.0 to 2.5]
  Swelling: Moderate | 2.9 [1.5 to 4.9] | 0.4 [0.0 to 2.5]
  Swelling: Severe | 0.2 [0.0 to 1.2] | 0 [0.0 to 1.6]

2. Primary Outcome: SSA: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, vomiting, nausea, diarrhea, muscle pain and joint pain. These were recorded by participants in an e-diary. Fever defined as oral temperature >=38.0 degrees Celsius (deg C) and categorized as mild: >=38.0 to 38.4 deg C, moderate: >38.4 to 38.9 deg C and severe: >38.9 to 40.0 deg C. Vomiting categorized as mild: 1-2 times in 24 hours (h); moderate: >2 times in 24h; severe: required intravenous (IV) hydration. Diarrhea categorized as mild: 2-3 loose stools in 24h; moderate: 4-5 loose stools in 24h; severe: 6 or more loose stools in 24h. Headache, fatigue, nausea, muscle pain and joint pain were categorized as mild: didn't interfere with activity; moderate: some interference with activity; severe: prevented daily routine activity.
Time Frame: Within 7 Days after Vaccination (Vaccination on Day 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: RSVpreF | SSA: Placebo
Number analyzed (Participants) | 451 | 225
Percentage of participants
  Fever: 38.0°C to 38.4°C | 0.4 [0.1 to 1.6] | 0.4 [0.0 to 2.5]
  Fever: >38.4°C to 38.9°C | 1.1 [0.4 to 2.6] | 0.9 [0.1 to 3.2]
  Fever: >38.9°C to 40.0°C | 0 [0.0 to 0.8] | 0 [0.0 to 1.6]
  Fatigue: Mild | 18.2 [14.7 to 22.1] | 22.2 [17.0 to 28.2]
  Fatigue: Moderate | 18.2 [14.7 to 22.1] | 15.6 [11.1 to 21.0]
  Fatigue: Severe | 0.9 [0.2 to 2.3] | 0.4 [0.0 to 2.5]
  Headache: Mild | 20.8 [17.2 to 24.9] | 18.7 [13.8 to 24.4]
  Headache: Moderate | 7.3 [5.1 to 10.1] | 11.6 [7.7 to 16.5]
  Headache: Severe | 0.2 [0.0 to 1.2] | 0 [0.0 to 1.6]
  Muscle Pain: Mild | 15.7 [12.5 to 19.4] | 9.8 [6.2 to 14.4]
  Muscle Pain: Moderate | 8.6 [6.2 to 11.6] | 6.2 [3.4 to 10.2]
  Muscle Pain: Severe | 0 [0.0 to 0.8] | 0 [0.0 to 1.6]
  Joint Pain: Mild | 7.1 [4.9 to 9.9] | 4.0 [1.8 to 7.5]
  Joint Pain: Moderate | 5.1 [3.3 to 7.6] | 6.2 [3.4 to 10.2]
  Joint Pain: Severe | 0.2 [0.0 to 1.2] | 0 [0.0 to 1.6]
  Nausea: Mild | 9.3 [6.8 to 12.4] | 8.9 [5.5 to 13.4]
  Nausea: Moderate | 2.4 [1.2 to 4.3] | 0.9 [0.1 to 3.2]
  Nausea: Severe | 0 [0.0 to 0.8] | 0.4 [0.0 to 2.5]
  Vomiting: Mild | 1.6 [0.6 to 3.2] | 0.4 [0.0 to 2.5]
  Vomiting: Moderate | 0.4 [0.1 to 1.6] | 0.9 [0.1 to 3.2]
  Vomiting: Severe | 0 [0.0 to 0.8] | 0 [0.0 to 1.6]
  Diarrhea: Mild | 11.1 [8.3 to 14.4] | 12.4 [8.4 to 17.5]
  Diarrhea: Moderate | 3.1 [1.7 to 5.2] | 3.6 [1.5 to 6.9]
  Diarrhea: Severe | 0.7 [0.1 to 1.9] | 0.9 [0.1 to 3.2]

3. Primary Outcome: SSA: Percentage of Participants With Adverse Events (AEs) From Vaccination Through 1 Month After Vaccination
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were included. AEs included both serious and all non-serious adverse events.
Time Frame: Within 1 Month after Vaccination (Vaccination on Day 1)
Population: Safety population included all enrolled participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: RSVpreF | SSA: Placebo
Number analyzed (Participants) | 453 | 225
Percentage of participants | 7.1 [4.9 to 9.8] | 7.6 [4.5 to 11.8]

4. Primary Outcome: SSA: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Vaccination Throughout the Study
Description: A NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects. Newly diagnosed chronic medical condition did not include illnesses considered to be temporary conditions.
Time Frame: Within 6 Months after Vaccination (Vaccination on Day 1)
Population: Safety population included all enrolled participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: RSVpreF | SSA: Placebo
Number analyzed (Participants) | 453 | 225
Percentage of participants | 0.7 [0.1 to 1.9] | 2.2 [0.7 to 5.1]

5. Primary Outcome: SSA: Percentage of Participants With Serious Adverse Events (SAEs) Throughout the Study
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event were included in this outcome measure.
Time Frame: Within 6 Months after Vaccination (Vaccination on Day 1)
Population: Safety population included all enrolled participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: RSVpreF | SSA: Placebo
Number analyzed (Participants) | 453 | 225
Percentage of participants | 1.1 [0.4 to 2.6] | 3.1 [1.3 to 6.3]

6. Primary Outcome: SSA: Geometric Mean Ratio (GMR) Estimated by Ratio of the Geometric Mean Titers (GMTs) at 1 Month After Vaccination in Study C3671023 Participants Compared to Study C3671013 Adults >= 60 Years
Description: In this outcome measure, GMTs for RSV A and RSV B neutralizing titers (NTs) are reported. In statistical section, GMT ratio estimated by the ratio of the GMTs for RSV A and RSV B serum NTs at 1 month after vaccination with RSVpreF in current study C3671023 participants to that in study C3671013 adults >=60 years of age, is reported. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student t distribution).
Time Frame: At 1 Month after Vaccination (Vaccination on Day 1)
Population: C3671023: Evaluable immunogenicity population: participants eligible for SSA; received study interventions (RSVpreF or placebo) to which they were randomized; had 1-month postvaccination blood collection 27-42 days after vaccination; had at least 1 valid and determinate assay result 1 month after vaccination; had no major protocol violations from vaccination up to 1-month postvaccination blood draw. C3671013: Immunogenicity subset. "Number Analyzed" = participants evaluable for specified rows.
Measure: Least Squares Mean (95% Confidence Interval); unit: Titer
Groups:
- C3671023 SSA: RSVpreF: Participants aged >=18 to <60 years received RSVpreF 120 mcg intramuscularly on Day 1 of SSA.
- C3671013: RSVpreF, >=60 Years: Participants aged >=60 years who were vaccinated with RSVpreF 120 mcg in C3671013 study are included. Only the relevant historical data from these participants is utilized, they are not enrolled in the present study.
Arm/Group | C3671023 SSA: RSVpreF | C3671013: RSVpreF, >=60 Years
Number analyzed (Participants) | 437 | 408
Titer
  RSV A: number analyzed (Participants) | 435 | 408
  RSV A | 41097 [37986.1 to 44463.4] | 26225 [24143.1 to 28485.7]
  RSV B | 37416 [34277.9 to 40842.0] | 24680 [22504.3 to 27065.4]
Statistical Analysis 1: Comparison: C3671023 SSA: RSVpreF vs C3671013: RSVpreF, >=60 Years; Test type: Non-Inferiority — Noninferiority was declared if both the null hypothesis of GMR and the null hypothesis of difference in seroresponse rates were rejected for both RSV A and RSV B serum NTs, with a type I error (2-sided) of 5%; GMR = 1.57, 95% CI 2-sided [1.396 to 1.759] — GMRs (ratio of GMTs from C3671023 SSA to C3671013 immunogenicity subset), 2-sided CI were calculated by exponentiating difference in LS means, corresponding CIs based on regression model. Data reported here is for RSV A
Statistical Analysis 2: Comparison: C3671023 SSA: RSVpreF vs C3671013: RSVpreF, >=60 Years; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; GMR = 1.52, 95% CI 2-sided [1.333 to 1.725] — GMRs (ratio of GMTs from C3671023 SSA to C3671013 immunogenicity subset), 2-sided CI were calculated by exponentiating difference in LS means, corresponding CIs based on regression model. Data reported here is for RSV B

7. Primary Outcome: SSA: Percentage of Participants With Seroresponse Rate and Difference in Seroresponse Rates of RSV A and RSV B Serum NTs at 1 Month After Vaccination for Participants in Study C3671023 and C3671013 Adults >= 60 Years
Description: Seroresponse was defined as achieving a >=4-fold rise from baseline (before vaccination), if the baseline measurement was above the lower limit of quantitation (LLOQ). If the baseline measurement was below the LLOQ, a postvaccination assay result >=4* LLOQ was considered a seroresponse.
Time Frame: At 1 Month after Vaccination (Vaccination on Day 1)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C3671023 SSA: RSVpreF | C3671013: RSVpreF, >=60 Years
Number analyzed (Participants) | 437 | 408
Percentage of participants
  RSV A: number analyzed (Participants) | 435 | 408
  RSV A | 93.1 [90.3 to 95.3] | 88.0 [84.4 to 91.0]
  RSV B | 93.4 [90.6 to 95.5] | 85.0 [81.2 to 88.4]
Statistical Analysis 1: Comparison: C3671023 SSA: RSVpreF vs C3671013: RSVpreF, >=60 Years; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Difference in percentage = 5.1, 95% CI 2-sided [1.2 to 9.2] — Difference (C3671023 SSA, compared to C3671013 immunogenicity subset) in proportions, expressed as a percentage; 95% CIs for percentage difference were calculated using exact method based on Miettinen and Nurminen. Data reported here is for RSV A
Statistical Analysis 2: Comparison: C3671023 SSA: RSVpreF vs C3671013: RSVpreF, >=60 Years; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Difference in percentage = 8.3, 95% CI 2-sided [4.2 to 12.6] — Difference (C3671023 SSA, compared to C3671013 immunogenicity subset) in proportions, expressed as a percentage; 95% CIs for percentage difference were calculated using exact method based on Miettinen and Nurminen. Data reported here is for RSV B

8. Primary Outcome: SSB: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions included pain at injection site, redness and swelling, recorded by participants in an e-diary. Pain at injection site was graded as mild: did not interfere with activity; moderate: interfered with activity and severe: prevented daily activity. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 cm. Redness and swelling were graded as mild: > 2.0 cm to 5.0 cm; moderate: > 5.0 cm to 10.0 cm and severe: > 10 cm.
Time Frame: Within 7 Days after Vaccination 1 (Vaccination 1 on Day 1)
Population: E-diary safety population included all participants who received the first dose of RSVpreF and had at least 1 day of e-diary data transferred during the Dose 1 e-diary collection period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 96 | 107
Percentage of participants
  Pain at injection site: Mild | 25.0 [16.7 to 34.9] | 16.8 [10.3 to 25.3]
  Pain at injection site: Moderate | 1.0 [0.0 to 5.7] | 0 [0.0 to 3.4]
  Pain at injection site: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Redness: Mild | 5.2 [1.7 to 11.7] | 1.9 [0.2 to 6.6]
  Redness: Moderate | 1.0 [0.0 to 5.7] | 1.9 [0.2 to 6.6]
  Redness: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Swelling: Mild | 6.3 [2.3 to 13.1] | 0.9 [0.0 to 5.1]
  Swelling: Moderate | 2.1 [0.3 to 7.3] | 1.9 [0.2 to 6.6]
  Swelling: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]

9. Primary Outcome: SSB: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions included pain at injection site, redness and swelling, recorded by participants in an e-diary. Pain at injection site was graded as mild: did not interfere with activity; moderate: interfered with activity and severe: prevented daily activity. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit = 0.5 cm. Redness and swelling were graded as mild: >2.0 cm to 5.0 cm; moderate: >5.0 cm to 10.0 cm and severe: >10 cm.
Time Frame: Within 7 Days after Vaccination 2 (Vaccination 2: 1-month post-vaccination 1 on Day 1)
Population: E-diary safety population included all participants who received 2 doses of RSVpreF and had at least 1 day of e-diary data transferred during the Dose 2 e-diary collection period. Here, 'Overall Number of Participants Analyzed' (N)= participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 94 | 105
Percentage of participants
  Pain at injection site: Mild | 42.6 [32.4 to 53.2] | 29.5 [21.0 to 39.2]
  Pain at injection site: Moderate | 4.3 [1.2 to 10.5] | 1.9 [0.2 to 6.7]
  Pain at injection site: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Redness: Mild | 2.1 [0.3 to 7.5] | 1.9 [0.2 to 6.7]
  Redness: Moderate: number analyzed (Participants) | 94 | 104
  Redness: Moderate | 0 [0.0 to 3.8] | 1.9 [0.2 to 6.7]
  Redness: Severe: number analyzed (Participants) | 94 | 104
  Redness: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Swelling: Mild | 2.1 [0.3 to 7.5] | 3.8 [1.0 to 9.5]
  Swelling: Moderate | 1.1 [0.0 to 5.8] | 5.7 [2.1 to 12.0]
  Swelling: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]

10. Primary Outcome: SSB: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: as for outcome 2
Time Frame: Within 7 Days after Vaccination 1 (Vaccination 1 on Day 1)
Population: as for outcome 8
Measure: Number (96% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 96 | 107
Percentage of participants
  Fever: 38.0°C to 38.4°C | 1.0 [0.0 to 5.7] | 0.9 [0.0 to 5.1]
  Fever: >38.4°C to 38.9°C | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Fever: >38.9°C to 40.0°C | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Fatigue: Mild | 20.8 [13.2 to 30.3] | 19.6 [12.6 to 28.4]
  Fatigue: Moderate | 16.7 [9.8 to 25.6] | 22.4 [14.9 to 31.5]
  Fatigue: Severe | 2.1 [0.3 to 7.3] | 2.8 [0.6 to 8.0]
  Headache: Mild | 29.2 [20.3 to 39.3] | 15.0 [8.8 to 23.1]
  Headache: Moderate | 9.4 [4.4 to 17.1] | 6.5 [2.7 to 13.0]
  Headache: Severe | 0 [0.0 to 3.8] | 0.9 [0.0 to 5.1]
  Vomiting: Mild | 4.2 [1.1 to 10.3] | 0.9 [0.0 to 5.1]
  Vomiting: Moderate | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Vomiting: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Nausea: Mild | 9.4 [4.4 to 17.1] | 3.7 [1.0 to 9.3]
  Nausea: Moderate | 3.1 [0.6 to 8.9] | 4.7 [1.5 to 10.6]
  Nausea: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Diarrhea: Mild | 15.6 [9.0 to 24.5] | 12.1 [6.6 to 19.9]
  Diarrhea: Moderate | 6.3 [2.3 to 13.1] | 5.6 [2.1 to 11.8]
  Diarrhea: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.4]
  Muscle Pain: Mild | 18.8 [11.5 to 28.0] | 13.1 [7.3 to 21.0]
  Muscle Pain: Moderate | 7.3 [3.0 to 14.4] | 5.6 [2.1 to 11.8]
  Muscle Pain: Severe | 0 [0.0 to 3.8] | 1.9 [0.2 to 6.6]
  Joint Pain: Mild | 10.4 [5.1 to 18.3] | 11.2 [5.9 to 18.8]
  Joint Pain: Moderate | 7.3 [3.0 to 14.4] | 8.4 [3.9 to 15.4]
  Joint Pain: Severe | 0 [0.0 to 3.8] | 1.9 [0.2 to 6.6]

11. Primary Outcome: SSB: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: as for outcome 2
Time Frame: Within 7 Days after Vaccination 2 (Vaccination 2: 1-month post-vaccination 1 on Day 1)
Population: E-diary safety population included all participants who received 2 doses of RSVpreF and had at least 1 day of e-diary data transferred during the Dose 2 e-diary collection period. Here, 'N'= participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 94 | 105
Percentage of participants
  Fever: 38.0°C to 38.4°C | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Fever: >38.4°C to 38.9°C | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Fever: >38.9°C to 40.0°C | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Fatigue: Mild | 19.1 [11.8 to 28.6] | 23.8 [16.0 to 33.1]
  Fatigue: Moderate | 18.1 [10.9 to 27.4] | 19.0 [12.0 to 27.9]
  Fatigue: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Headache: Mild | 13.8 [7.6 to 22.5] | 19.0 [12.0 to 27.9]
  Headache: Moderate | 10.6 [5.2 to 18.7] | 5.7 [2.1 to 12.0]
  Headache: Severe | 0 [0.0 to 3.8] | 1.0 [0.0 to 5.2]
  Vomiting: Mild | 2.1 [0.3 to 7.5] | 1.0 [0.0 to 5.2]
  Vomiting: Moderate | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Vomiting: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Nausea: Mild | 5.3 [1.7 to 12.0] | 5.7 [2.1 to 12.0]
  Nausea: Moderate | 1.1 [0.0 to 5.8] | 1.0 [0.0 to 5.2]
  Nausea: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Diarrhea: Mild | 6.4 [2.4 to 13.4] | 10.5 [5.3 to 18.0]
  Diarrhea: Moderate | 5.3 [1.7 to 12.0] | 2.9 [0.6 to 8.1]
  Diarrhea: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Muscle Pain: Mild | 16.0 [9.2 to 25.0] | 15.2 [9.0 to 23.6]
  Muscle Pain: Moderate | 3.2 [0.7 to 9.0] | 8.6 [4.0 to 15.6]
  Muscle Pain: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]
  Joint Pain: Mild | 8.5 [3.7 to 16.1] | 12.4 [6.8 to 20.2]
  Joint Pain: Moderate | 3.2 [0.7 to 9.0] | 4.8 [1.6 to 10.8]
  Joint Pain: Severe | 0 [0.0 to 3.8] | 0 [0.0 to 3.5]

12. Primary Outcome: SSB: Percentage of Participants With AEs From Vaccination 1 Through 1 Month After Vaccination 2
Description: as for outcome 3
Time Frame: From Vaccination 1 (on Day 1) through 1 month after Vaccination 2 (1 month after Vaccination 1) [approximately up to maximum of 2 months]
Population: Safety population included all enrolled participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 96 | 107
Percentage of participants | 13.5 [7.4 to 22.0] | 22.4 [14.9 to 31.5]

13. Primary Outcome: SSB: Percentage of Participants With NDCMCs From Vaccination Throughout the Study
Description: as for outcome 4
Time Frame: From Vaccination 1 (on Day 1) through 6 months after Vaccination 2 (1 month after Vaccination 1) [approximately up to maximum of 7 months]
Population: Safety population included all enrolled participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 96 | 107
Percentage of participants | 2.1 [0.3 to 7.3] | 6.5 [2.7 to 13.0]

14. Primary Outcome: SSB: Percentage of Participants With SAEs Throughout the Study
Description: as for outcome 5
Time Frame: as for outcome 13
Population: Safety population included all enrolled participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 96 | 107
Percentage of participants | 7.3 [3.0 to 14.4] | 14.0 [8.1 to 22.1]

15. Primary Outcome: SSB: GMT of NT for RSV A and RSV B Before Vaccination 1
Description: GMT of RSV A and RSV B before vaccination were reported in this outcome measure. Assay results below the lower limit of quantification (LLOQ) were set to 0.5*LLOQ. GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution).
Time Frame: Before Vaccination 1 (on Day 1)
Population: Evaluable immunogenicity population included all eligible participants for SSB who received 2 dose of RSVpreF; (blood collected for 1 month after last dose to be 27-42 days after second dose of RSVpreF; had at least 1 valid, determinate assay result 1 month after vaccination (1 month after second dose of RSVpreF); had no major protocol violations from vaccination through 1-month postvaccination blood draw (1 month after second dose of RSVpreF).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 90 | 98
Titer
  RSV A | 2943 [2417.9 to 3580.9] | 3289 [2735.1 to 3954.1]
  RSV B | 2584 [2120.6 to 3147.9] | 2992 [2416.5 to 3704.1]

16. Primary Outcome: SSB: GMT of NT for RSV A and RSV B 1 Month After Vaccination 1
Description: as for outcome 15
Time Frame: 1 Month After Vaccination 1 (on Day 1)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 90 | 98
Titer
  RSV A | 26173 [19937.1 to 34359.2] | 26075 [20513.1 to 33144.1]
  RSV B | 24701 [18300.5 to 33340.1] | 25384 [19749.5 to 32626.2]

17. Primary Outcome: SSB: GMT of NT for RSV A and RSV B 1 Month After Vaccination 2
Description: as for outcome 15
Time Frame: 1 Month After Vaccination 2 (1-month post Vaccination 1)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 90 | 98
Titer
  RSV A | 21910 [17308.8 to 27733.3] | 25159 [20085.1 to 31515.2]
  RSV B | 20936 [16154.0 to 27134.4] | 22774 [18016.7 to 28788.3]

18. Secondary Outcome: SSB: Geometric Mean Fold Rise (GMFR) of NTs for RSV A and RSV B From Vaccination 1 to 1 Month Post-Vaccination 1
Description: GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution).
Time Frame: At 1 Month After Vaccination 1 (on Day 1) to 1 Month Post-Vaccination 1
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 90 | 98
Fold rise
  RSV A | 8.8 [6.76 to 11.53] | 7.9 [6.21 to 10.13]
  RSV B | 9.6 [7.31 to 12.51] | 8.5 [6.70 to 10.75]

19. Secondary Outcome: SSB: GMFR of NTs for RSV A and RSV B From Vaccination 1 to 1 Month Post-Vaccination 2
Description: as for outcome 18
Time Frame: At 1 Month After Vaccination 1 (on Day 1) to 1 Month Post-Vaccination 2
Population: Evaluable immunogenicity population was analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
Number analyzed (Participants) | 90 | 98
Fold rise
  RSV A | 7.4 [5.88 to 9.29] | 7.7 [6.11 to 9.58]
  RSV B | 8.1 [6.45 to 10.18] | 7.6 [6.06 to 9.57]

20. Secondary Outcome: SSA: GMT of NTs for RSV A and RSV B Before Vaccination and 1 Month After Vaccination
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution).
Time Frame: SSA: Before Vaccination (on Day 1) and 1 Month After Vaccination
Population: Evaluable immunogenicity population=participants who met following criteria:(i)eligible for Substudy A;(ii)received study interventions (RSVpreF or placebo)to which they were randomized;(iii)had 1-month postvaccination blood collected 27-42days after vaccination;(iv) had at least 1 valid,determinate assay result 1month after vaccination;(v)had no major protocol violations from vaccination through 1-month postvaccination blood draw. Here,'Number Analyzed'=participants evaluable at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSA: RSVpreF | SSA: Placebo
Number analyzed (Participants) | 437 | 217
Titer
  RSV A: Before Vaccination: number analyzed (Participants) | 436 | 217
  RSV A: Before Vaccination | 2388 [2207.7 to 2583.3] | 2797 [2516.8 to 3108.9]
  RSV A: 1 month after vaccination: number analyzed (Participants) | 436 | 217
  RSV A: 1 month after vaccination | 41595 [38416.6 to 45037.5] | 2660 [2395.2 to 2953.9]
  RSV B: Before Vaccination | 2075 [1899.7 to 2265.4] | 2230 [1988.6 to 2501.6]
  RSV B: 1 month after vaccination | 38450 [35187.5 to 42014.7] | 2135 [1905.9 to 2391.3]

21. Secondary Outcome: SSA: GMFR of NTs for RSV A and RSV B From Before Vaccination to 1 Month After Vaccination
Description: as for outcome 18
Time Frame: SSA: Before Vaccination (on Day 1) and 1 Month After Vaccination
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSA: RSVpreF | SSA: Placebo
Number analyzed (Participants) | 437 | 217
Fold rise
  RSV A: number analyzed (Participants) | 435 | 217
  RSV A | 17.5 [15.88 to 19.21] | 1.0 [0.90 to 1.00]
  RSV B | 18.5 [16.76 to 20.43] | 1.0 [0.91 to 1.01]

ADVERSE EVENTS:
Time Frame: SSA- LR/SE: Within 7Days after Vaccination (Vacc on Day1);AEs: Within 1 Month (M) after Vacc (Vacc on Day1), including any events reported up to 6 months; SAEs: Any events reported up to 6 months; SSB- LR/SE: Within 7 Days after Vacc1 (Day1 of SSB) Within 7 Days after Vacc 2 (second dose on 1M post-vacc.1); AEs: From Vacc 1 (on Day1) through 1M after Vacc 2 (1M after Vacc1) [approximately up to maximum of 2M], including any events reported up to 7 months; SAEs: any events reported up to 7 months
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population included all enrolled participants who received the study intervention.
Arm/Group | SSA: RSVpreF | SSA: Placebo | SSB: RSVpreF, >= 18 to < 60 Years | SSB: RSVpreF, >= 60 Years
All-Cause Mortality (participants affected / at risk) | 1/453 | 0/225 | 0/96 | 0/107
Serious Adverse Events (participants affected / at risk) | 5/453 | 7/225 | 7/96 | 15/107
Other Adverse Events (participants affected / at risk) | 301/453 | 135/225 | 73/96 | 92/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SSA: RSVpreF (N=453) | SSA: Placebo (N=225) | SSB: RSVpreF, >= 18 to < 60 Years (N=96) | SSB: RSVpreF, >= 60 Years (N=107)
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
SARS-CoV-2 sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SSA: RSVpreF (N=453) | SSA: Placebo (N=225) | SSB: RSVpreF, >= 18 to < 60 Years (N=96) | SSB: RSVpreF, >= 60 Years (N=107)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Epiretinal membrane (Eye disorders) | 1 | 0 | 0 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Fatigue (FATIGUE) (General disorders) | 168 | 86 | 52 | 62
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 159 | 24 | 54 | 41
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (FEVER) (General disorders) | 7 | 3 | 1 | 1
Swelling (SWELLING) (General disorders) | 32 | 2 | 9 | 12
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 67 | 38 | 28 | 27
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (NAUSEA) (Gastrointestinal disorders) | 53 | 23 | 15 | 13
Vomiting (VOMITING) (Gastrointestinal disorders) | 9 | 3 | 5 | 2
Primary biliary cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 7 | 3 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 5
Urinary tract infection (Infections and infestations) | 1 | 4 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 4
Hepatobiliary procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 56 | 23 | 21 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 110 | 36 | 32 | 33
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (HEADACHE) (Nervous system disorders) | 128 | 68 | 42 | 38
Migraine (Nervous system disorders) | 0 | 1 | 3 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 27 | 1 | 7 | 8
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Physical assault (Social circumstances) | 1 | 0 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 3
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Computerised tomogram abnormal (Investigations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Vertebral artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT05842967/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT05842967/SAP_001.pdf